CLINICAL TRIAL: NCT03607461
Title: Traditional Home Health Physical Therapy Versus a Smartphone App for Patients Recovering From Total Knee Arthroplasty During the Home-bound Portion of Recovery: Study Protocol for a Randomized Controlled Trial
Brief Title: Using a Smartphone App to Aid in Functional Mobility Return Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lagniappe Physical Therapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4357
Record Dates: First submitted 2018-07-03; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Control group will consist of those who meet the inclusion criteria and have received traditional home health services following total knee arthroplasty (TKA). Intervention group participants who meet the inclusion criteria will receive a smartphone app instead of traditional home health services to aid in knee mobility recovery following TKA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone App Users (Experimental): Smartphone App Users will receive important information and prescriptive exercise via a smartphone app upon returning home from the hospital following total knee arthroplasty
  Interventions: Device: Smartphone App
- Home Health Users (Active Comparator): Home Health Users will have already undergone traditional home health physical therapy and/or skilled nursing for the purpose of comparing outcomes
  Interventions: Combination Product: Control Group

INTERVENTIONS:
Device: Smartphone App — Smartphone App Users will engage with the app at least daily and follow along with the prescriptive exercises as instructed.
  Arms: Smartphone App Users
Combination Product: Control Group — Home Health users will have received traditional home health physical therapy and skilled nursing services.
  Arms: Home Health Users

SUMMARY:
Traditional home health care for individuals recovering from unilateral TKA is expensive and provides a higher level of service than most individuals, aged 45 to 64, require. Use of smartphone technology has the potential to drive down costs while maintaining outcomes for this patient population. The proposed randomized controlled trial would determine the efficacy and proper dose-response of a smartphone app to reduce costs and maintain outcomes for the desired patient population compared to traditional home care.

DETAILED DESCRIPTION:
As of 2013, it was estimated that 4.0 million individuals in the U.S. were living with a TKA, representing 4.2% of the population fifty years of age or older (8). As of 2010, there were 81,489,445 people aged 45 to 64 in the U.S. (4), with a rate of 39.5 total knee arthroplasties per year per 10,000 individuals in that age group (3). Therefore, approximately 322,000 TKAs were performed in 2010 for those aged 45 to 64. A 2010 study from The Centers for Disease Control and Prevention found the average cost of home health care following TKA to be $3,709 per episode of care per patient (5). This results in nearly $1.2 billion dollars in U.S. healthcare spending in 2010 for home care following TKA for those aged 45 to 64. The reason for the high cost of home health care may be the state regulations governing home health care agencies. The Louisiana Department of Health and Hospitals states that 'skilled home health care,' found under the definition of 'home health agency' in the official Louisiana Home Health State Regulations, is to include skilled nursing and at least one of the following services: physical therapy, occupational therapy, speech therapy, medical social services, or home health aide services (9). These regulations place pressure, whether conscious or subconscious, on the home health agency to over utilize skilled nursing services for those patients aged 45 to 64 recovering from TKA. Skilled nursing home health care services for this particular patient population usually involves managing the patient's medications and providing wound care services. A cohort study by Bleijenberg et al published in the Journal of the American Geriatric Society in 2017 found that only 10.3% of adults aged 65 to 69, which is above the age cutoff for this prospective study, had difficulty with managing their medications (10). Also, in the author's clinical experience, it is rare for an orthopedic surgeon to allow any other clinician to manage post-operative dressing changes except those clinicians under the surgeon's direct supervision; though further research in this area would be helpful. Furthermore, utilization of TKA, and the home care cost associated with recovery from TKA, is on the rise. As of 2009, the number of primary TKAs performed annually in the U.S. among all age groups exceeded 620,000 procedures, which is more than doubled when compared to the previous decade (7). Smartphones and other technologies may provide a solution to the rising costs of home health care following TKA for those aged 45 to 64. Over the past decade, the smartphone has become an integral part of most people's lives. The latest Pew Research Data from February 2018 shows that 73% of individuals aged 50 to 64 own a smartphone (8). Smartphones would allow the patient to have direct multimedia access to a prescriptive exercise program designed by a licensed Physical Therapist without an in-person home visit, as well as to have communication directly with their Physical Therapist through secure in-app messaging or e-mail. The patient would benefit by having reduced intrusion in their home environment, convenient access to their Physical Therapist and their Physical Therapist's plan of care, and financial savings due to the elimination of home health care services following TKA. The Physical Therapist would benefit from the ability to quickly interact with the patient to mitigate any adverse events and to efficiently assist a greater number of patients compared to traditional home-based physical therapy. Third-party payors would benefit from drastically reduced home care costs for those recovering from TKA.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 45 to 64
* unilateral TKA
* subject discharged directly to home from the hospital

Exclusion Criteria:

* subject does not engage with the app within 24 hours of discharge from the hospital
* subject neglects to engage with the app over any 24-hour period during the study
* subject is readmitted to the hospital at any point during the home bound portion of their recovery

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Total Knee Range of Motion (ROM) change | Baseline and through study completion, usually 2 to 4 weeks
  Initial knee ROM will be taken within 48 hours of discharge home from hospital. Final knee ROM will be taken upon participant no longer being homebound and expressing readiness to begin outpatient physical therapy
Western Ontario and McMaster Universities Osteoarthritis Index (shortened version) | Baseline and through study completion, usually 2 to 4 weeks
  Questionnaire to be completed by participant at time of initial data collection described above. Final questionnaire also completed as described above

SECONDARY OUTCOMES:
Self-Reported App Engagement | Data collected at final assessment, usually 2 to 4 weeks
  Participant will self-report frequency of app engagement

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Rippetoe, DPT, Principal Investigator — Owner of Lagniappe Physical Therapy
Locations (1):
- Office, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make IPD available to other researchers

REFERENCES:
- [Result] Whitehouse SL, Lingard EA, Katz JN, Learmonth ID. Development and testing of a reduced WOMAC function scale. J Bone Joint Surg Br. 2003 Jul;85(5):706-11. PMID 12892194
- [Result] Abbott JH, Hobbs C, Gwynne-Jones D; MOA Trial Team. The ShortMAC: Minimum Important Change of a Reduced Version of the Western Ontario and McMaster Universities Osteoarthritis Index. J Orthop Sports Phys Ther. 2018 Feb;48(2):81-86. doi: 10.2519/jospt.2018.7676. Epub 2017 Oct 21. PMID 29056072
- [Result] Weinstein AM, Rome BN, Reichmann WM, Collins JE, Burbine SA, Thornhill TS, Wright J, Katz JN, Losina E. Estimating the burden of total knee replacement in the United States. J Bone Joint Surg Am. 2013 Mar 6;95(5):385-92. doi: 10.2106/JBJS.L.00206. PMID 23344005
- [Result] Losina E, Thornhill TS, Rome BN, Wright J, Katz JN. The dramatic increase in total knee replacement utilization rates in the United States cannot be fully explained by growth in population size and the obesity epidemic. J Bone Joint Surg Am. 2012 Feb 1;94(3):201-7. doi: 10.2106/JBJS.J.01958. PMID 22298051
- [Result] Bleijenberg N, Smith AK, Lee SJ, Cenzer IS, Boscardin JW, Covinsky KE. Difficulty Managing Medications and Finances in Older Adults: A 10-year Cohort Study. J Am Geriatr Soc. 2017 Jul;65(7):1455-1461. doi: 10.1111/jgs.14819. Epub 2017 Apr 5. PMID 28378345
- See also: Mobile Fact Sheet. Pew Research Center. 2018 Feb 5. — http://www.pewinternet.org/fact-sheet/mobile/
- See also: Louisiana Home Health State Regulations. Department of Health and Hospitals. Office of the Secretary. Bureau of Health Services Financing. Louisiana Register. Vol 27, No 12, 2001 Dec 20. Accessed online — http://ldh.la.gov/assets/medicaid/hss/docs/HHA_MLS_St_regs.pdf

DOCUMENTS (2):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT03607461/Prot_000.pdf
  • Informed Consent Form (2018-06-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03607461/ICF_001.pdf